CLINICAL TRIAL: NCT00717691
Title: Hallux Limitus Treated With Dynamic Splinting: A Randomized, Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008.003
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Hallux Limitus
Keywords: Hallux Limitus; Dynamic Splinting; Dynasplint
MeSH Terms: conditions — Hallux Limitus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Immediate fitting with dynamic splinting following diagnosis of hallux limitus.
  Interventions: Device: Metatarsophalangeal Extension Dynasplint System; Other: Standard of Care
- 2 (No Intervention): Control arm; patients only treated with standard of care following diagnosis of hallux limitus.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Metatarsophalangeal Extension Dynasplint System — Dynamic Splinting utilizes the protocols of Low-Load, Prolonged-Duration Stretch (LLPS) with calibrated, adjustable tension to increase the Total End Range Time (TERT) to reduce contracture. This unit is worn for 30 minutes, three times per day, (while seated or resting in bed) totaling 1.5 hours per day.
  Arms: 1
Other: Standard of Care — The current standard of care in treating Hallux Limitus will be given to all patients regardless of randomized categorization, and this includes: analgesic and nonsteroidal anti-inflammatory drugs (NSAIDs), orthotics with medial stiffness, and reduction of great toe movement in motions such as kneeling or squatting with the toes in an extended position.

SUMMARY:
The purpose of this study is to regain range of motion of the great toe with dynamic splinting which will help reduce great toe's pain and swelling.

DETAILED DESCRIPTION:
Determine the efficacy of dynamic splinting in treating patients with hallux limitus, in a randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Reduced flexibility in AROM of extension in the great toe
* Pain that is worsened by walking and/or squatting
* Impaired gait pattern

Exclusion Criteria:

* Metatarsal stress fracture
* Interdigital neuroma
* Sesamoid pathology
* Gout
* Metatarsalgia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change in Active Range of Motion of Hallux (great toe) Extension | Two Months

SECONDARY OUTCOMES:
Change in passive Range of Motion, Extension | same

CONTACTS AND LOCATIONS:
Overall Officials: Stanley R Kalish, DPM, FACFAS, Principal Investigator — Atlanta Foot and Leg Clinic; Buck Willis, PhD, Study Director — Dynasplint Systems, Inc.
Locations (2):
- United States (2):
  - Atlanta Foot and Leg Clinic, Jonesboro, Georgia
  - Ankle and Foot Centers, PC, Marietta, Georgia

REFERENCES:
- [Background] Goucher NR, Coughlin MJ. Hallux metatarsophalangeal joint arthrodesis using dome-shaped reamers and dorsal plate fixation: a prospective study. Foot Ankle Int. 2006 Nov;27(11):869-76. doi: 10.1177/107110070602701101. PMID 17144945
- [Background] Hockenbury RT. Forefoot problems in athletes. Med Sci Sports Exerc. 1999 Jul;31(7 Suppl):S448-58. doi: 10.1097/00005768-199907001-00006. PMID 10416546
- [Background] Willis B, John M. Dynamic Splinting Increases Flexion for Hallux Rigidus (Pilot Study). BioMechanics, 2007 Sept;14(9), pg49-53
- [Background] Brodsky JW, Baum BS, Pollo FE, Mehta H. Prospective gait analysis in patients with first metatarsophalangeal joint arthrodesis for hallux rigidus. Foot Ankle Int. 2007 Feb;28(2):162-5. doi: 10.3113/FAI.2007.0162. PMID 17296132
- [Background] Talarico LM, Vito GR, Goldstein L, Perler AD. Management of hallux limitus with distraction of the first metatarsophalangeal joint. J Am Podiatr Med Assoc. 2005 Mar-Apr;95(2):121-9. doi: 10.7547/0950121. PMID 15778469
- [Background] Payne C, Chuter V, Miller K. Sensitivity and specificity of the functional hallux limitus test to predict foot function. J Am Podiatr Med Assoc. 2002 May;92(5):269-71. doi: 10.7547/87507315-92-5-269. PMID 12015407
- [Background] Kennedy JG, Chow FY, Dines J, Gardner M, Bohne WH. Outcomes after interposition arthroplasty for treatment of hallux rigidus. Clin Orthop Relat Res. 2006 Apr;445:210-5. doi: 10.1097/01.blo.0000201166.82690.23. PMID 16467621
- [Background] DeFrino PF, Brodsky JW, Pollo FE, Crenshaw SJ, Beischer AD. First metatarsophalangeal arthrodesis: a clinical, pedobarographic and gait analysis study. Foot Ankle Int. 2002 Jun;23(6):496-502. doi: 10.1177/107110070202300605. PMID 12095117
- [Background] Canseco K, Long J, Marks R, Khazzam M, Harris G. Quantitative characterization of gait kinematics in patients with hallux rigidus using the Milwaukee foot model. J Orthop Res. 2008 Apr;26(4):419-27. doi: 10.1002/jor.20506. PMID 17972321
- [Background] Becher C, Kilger R, Thermann H. Results of cheilectomy and additional microfracture techniques for the treatment of hallux rigidus. Foot Ankle Surg. 2005;(10): 155-160
- [Background] Lau JT, Daniels TR. Outcomes following cheilectomy and interpositional arthroplasty in hallux rigidus. Foot Ankle Int. 2001 Jun;22(6):462-70. doi: 10.1177/107110070102200602. PMID 11475452
- [Background] Willis B. Dancers restore knee flexion through dynamic splinting. BioMechanics. 2008;Jan;15(1), pg49-54